CLINICAL TRIAL: NCT06724562
Title: An Observational Study of IL1 Inhibition for Blocking ACVR1-Induced Flare Activity and Heterotopic Ossification in Fibrodysplasia Ossificans Progressiva (FOP)
Brief Title: An Observational Pre-post Study to Observe if the Off Label Use of Anti-IL1 Therapies, Such as Anakinra or Canakinumab, Can Block ACVR1-induced Flare Activity and Heterotopic Ossification in FOP
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 23-40055; R01AR083628 (NIH)
Record Dates: First submitted 2024-11-27; First posted 2024-12-09 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Fibrodysplasia Ossificans Progressiva (FOP)
Keywords: heterotopic ossification; canakinumab; anakinra; FOP
MeSH Terms: conditions — Myositis Ossificans; Ossification, Heterotopic | interventions — canakinumab; Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for DNA, cell isolation, biochemistry, and cytokine analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Anti-IL1 Observational Arm: FOP patients that are beginning treatment with Anti-IL1 Therapy
  Interventions: Other: Anti-IL1 Therapy
- Optional Non-Treatment Observational Arm: FOP patients unable to obtain Anti-IL1 therapy
- "On Treatment" Observational Arm: FOP patients that are already using Anti-IL1 therapy

INTERVENTIONS:
Other: Anti-IL1 Therapy — Anti-IL1 is a rescue therapy for FOP patients that is hypothesized to reduce flare activity and subsequent ossification in these patients
  Other Names: Canakinumab; Anakinra
  Groups: Anti-IL1 Observational Arm

SUMMARY:
This is an observational pre-post study to observe if the off label use of anti-IL1 therapies, such as anakinra or canakinumab, can block ACVR1-induced flare activity and heterotopic ossification in FOP. It will also generate key tools and preliminary data that are needed to design a future Phase II study.

This study specifically focuses on patients with severe FOP who are being considered by their medical team for rescue therapy with anti-IL1 therapy. Preliminary data suggests patients experience significant decreases in flare frequency when taking anti-IL1 therapy, but other measures of efficacy remain unassessed, such as changes in heterotopic ossification formation, changes in pain medication use, and changes in functionality.

DETAILED DESCRIPTION:
The investigators will perform an observational study on patients with FOP who have decided, along with their primary medical team, to start anti-IL1 therapy with either anakinra or canakinumab due to intractable or unusually severe FOP disease progression. The investigators will study 11 subjects aged 6-30 years old, with a self-reported flare frequency of at least 4 flares/year [2 times above the average reported FOP population flare frequency of 2 flares/year] or with an intractable flare that has lasted greater than 1 month. Subjects will begin an observational period during the medication prescription and insurance approval process and will then be followed for up to 1 year after treatment has been initiated by the medical management team. Low-dose whole-body CT (WBCT) imaging, bloodwork, patient-reported outcomes, pain, and flare activity will be assessed during this study. In addition, patients who are currently on anti-IL1 therapy will be enrolled in a separate observation-only arm to collect historical data related to their experiences on therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical presentation consistent with FOP and a genetic diagnosis of classical FOP (ACVR1R206H variant) (2), male or female aged 6-30 years old.
* Patients with unusually severe FOP disease activity. This will be determined by FOP flare frequency of >4 flares per year, which is 2 times higher than the reported average in prior FOP studies ; or by a persistent flare that has failed to resolve after 1 month of standard-of-care therapy.
* Patients whose primary medical team has decided that rescue therapy with an anti-IL1 medication should be initiated. Once the primary medical team has decided that anti-IL1 therapy should be pursued, the subject will be told about this clinical-observational study and enrolled in the pre-treatment phase while access to the anti-IL1 therapy is being obtained by the clinical management team.
* Ability to participate in all assessments, including blood draws, radiology assessments, and travel. Age 6 is chosen as the lower limit to avoid the need for anesthesia for whole body CT in younger subjects.
* No history of unexplained infections, known autoimmune disease, or contraindication to anti-IL1 therapy.
* Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
* Inability to travel to site for assessments
* Pre-existing autoimmune or autoinflammatory disease (aside from FOP)
* Inability to tolerate assessments (such as phlebotomy)
* Unexplained infections
* Current participation in an interventional trial, or study of a potentially disease modifying medication
* Inability to take medications as prescribed by managing physician

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects with a diagnosis of FOP who meet the inclusion and exclusion criteria will be eligible for participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of flares that a patient experiences. | 1 year
  Surveys will be used to track the number of clinical flares that a patient experiences before and during treatment with anti-IL1 therapy.

SECONDARY OUTCOMES:
Change in new heterotopic ossification bone formation over time | 1 year
  Low dose whole body CT (WBCT) without the head, will be used to create detailed images of the skeletal system. The images will be used to measure new HO bone formation from baseline.
Changes in blood inflammatory cytokine levels with anti-IL1 therapy | 1 year
  Blood samples will be taken to measure changes in the inflammatory cytokines present in the blood over time, and if this changes with anti-IL1 treatment.
Change in patient mobility | 1 year
  The Cumulative Analog Joint Involvement Scale (CAJIS) will be used to assess 15 major joints for their mobility. This will be compared from baseline vs. 1 year of anti-IL1 treatment.
Number of participants with treatment emergent adverse events (TEAEs) | 1 year
  The number of participants with adverse events (ie adverse events not at baseline) will be collected during the treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Hsiao, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient data will be deidentified and shared following NIH policies for aggregate and individual level data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 2 years of the end of the study.

REFERENCES:
- [Background] Haviv R, Zeitlin L, Moshe V, Ziv A, Rabinowicz N, De Benedetti F, Prencipe G, Matteo V, De Cunto CL, Hsiao EC, Uziel Y. Long-term use of interleukin-1 inhibitors reduce flare activity in patients with fibrodysplasia ossificans progressiva. Rheumatology (Oxford). 2024 Sep 1;63(9):2597-2604. doi: 10.1093/rheumatology/keae255. PMID 38733591
- [Background] Haviv R, Moshe V, De Benedetti F, Prencipe G, Rabinowicz N, Uziel Y. Is fibrodysplasia ossificans progressiva an interleukin-1 driven auto-inflammatory syndrome? Pediatr Rheumatol Online J. 2019 Dec 21;17(1):84. doi: 10.1186/s12969-019-0386-6. PMID 31864380